CLINICAL TRIAL: NCT03524053
Title: Mediator Release During Exercise-induced Bronchoconstriction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brunel University (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Hannah Marshall, PhD Research Student, Brunel University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 8666
Record Dates: First submitted 2018-04-20; First posted 2018-05-14 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Exercise Induced Asthma
MeSH Terms: conditions — Asthma, Exercise-Induced

STUDY DESIGN:
Intervention Model Description: Patients will undertake 3 separate conditions in a randomised order.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercise induced bronchoconstriction (Experimental): An exercise challenge will then be performed according to international guidelines. The exercise will consist of 8 minutes of cycling on a cycle ergometer while breathing medical grade dry air from a reservoir (Douglas bag) via a two-way non-rebreathing valve. The workload will be increased progressively over the first 2 minutes, and will then be maintained for 6 minutes at a target workload (in Watts) of [53.76 * measured forced expiratory volume in 1 sec (FEV1)-11.07].
  Interventions: Other: Exercise induced bronchoconstriction
- Inhibited EIB (Active Comparator): An exercise challenge will then be performed according to international guidelines. The exercise will consist of 8 minutes of cycling on a cycle ergometer while warm-humid air from a reservoir (Douglas bag) via a two-way non-rebreathing valve. The workload will be increased progressively over the first 2 minutes, and will then be maintained for 6 minutes at a target workload (in Watts) of [53.76 * measured forced expiratory volume in 1 sec (FEV1)-11.07].
  Interventions: Other: Inhibited EIB
- Control (No Intervention): Participants will attend the laboratory but no exercise trial will be performed.

INTERVENTIONS:
Other: Exercise induced bronchoconstriction — Participants will exercise whilst inhaling dry-air, this is known to exacerbate the bronchoconstrictive response.
  Other Names: Induced bronchoconstriction
  Arms: Exercise induced bronchoconstriction
Other: Inhibited EIB — Participants will perform the exercise-test whilst inhaling warm-humid air. This is known to inhibit the EIB response and will provide a direct comparison group for the EIB condition.
  Other Names: Exercise-control
  Arms: Inhibited EIB

SUMMARY:
This study will compare the inflammatory response in induced vs inhibited exercise induced bronchoconstriction (EIB) in patients with a medical diagnosis of asthma/EIB. Urinary and plasma samples will be analysed to compare the mediator release in each condition, alongside changes in lung function.

DETAILED DESCRIPTION:
Exercise induced-bronchoconstriction (EIB) is a transient narrowing of the airways that occurs during or shortly after strenuous exercise. The prevalence of EIB in asthmatic patients is estimated around 30-50%, but EIB can also occur in individuals without asthma (especially children, army recruit forces, and elite athletes). Controversy remains about the causative mediators in the bronchoconstrictive response. Technological advancement in mass spectrometry has opened new avenues in the quantitative measurement of small endogenous metabolites in biological fluids (including urine and blood), which may provide insights into the pathophysiology of EIB and direct future therapeutic targets.

Utilising novel techniques in the analysis of inflammatory mediators in urine and blood, this study aims to conduct the most comprehensive analysis of mediator release during EIB to date.

Participants will attend a screening visit during which they will complete an exercise challenge (to determine the presence of EIB). A skin prick test will also be conducted to establish the atopic status of the participants. Following the screening visit, patients with EIB will be invited to complete a randomised cross-over study, where they will perform two further exercise challenges on separate days: one while inhaling temperate dry air, and one while inhaling hot humid air (the latter is known to inhibit EIB). Lung function and breathing discomfort will be recorded, and urine and blood samples will be collected, before and at various time points after exercise. As a control condition, participants will also attend one visit during which no exercise will be performed.

Participants aged 18-50yr, with diagnosed asthma and/or EIB, will be included in the study. 12 participants will complete 4 visits (lasting between 90 min and 4.5h). The study will take place on Brunel University London campus, Uxbridge. Urine and blood samples will be sent to the Karolinska Institutet, Stockholm, Sweden for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand the study instructions
* Willing and able to give informed consent
* Aged 18-50yr
* Physician-diagnosed asthma and/or EIB
* Participants that demonstrate EIB at the screening visit (i.e., those who have a fall in FEV1 20% to 50%) will be eligible for the full study.

Exclusion Criteria:

* Any chronic medical condition other than asthma or EIB
* Baseline FEV1 <70% predicted
* Exacerbation of asthma or respiratory infection within the last 4 wk
* Individuals who have varied their inhaled corticosteroid medication within the last 4 wk
* History of anaphylaxis
* Current smokers
* Pregnancy
* History of cardiovascular disease
* Injury that would prevent exercise on a cycle ergometer
* Medical contraindication to perform strenuous exercise
* Required oral corticosteroids in the past 3 months
* Any blood borne disease

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Changes in the concentration of inflammatory mediator metabolites in urine | Urine sample will be collected 45 minutes and immediately prior to the exercise challenges (or controlled resting period) and at 45, 90, 135 and 180 minutes post-exercise.
  Concentration of metabolites of prostaglandin-D2, Cysteinyl-Leukotrienes, prostaglandin-E2, prostacyclin, thromboxane and isoprostanes will be expressed as pg per mmol of creatinine.

SECONDARY OUTCOMES:
Changes in the concentration of inflammatory mediator metabolites in blood plasma | Urine sample will be collected 45 minutes and immediately prior to the exercise challenges (or controlled resting period) and at 45, 90, 135 and 180 minutes post-exercise.
  Concentration of tryptase and pro-inflammatory cytokines measured from blood plasma samples.
Forced vital capacity (FVC) manoeuvres using spirometry | Spirometry will be performed 45 minutes and immediately prior to the exercise challenges (or controlled resting period) and at 45, 90, 135 and 180 minutes post-exercise.
  Forced expiratory volume in one second (FEV1) measured in litres will be used to determine the severity of EIB from baseline to post-exercise challenge.
Breathing rate | Continuous recording throughout 8-min exercise test using the online breath-by-breath analysis system.
  Breathing rate (breaths per minute) will be recorded throughout exercise to control intensity between trials.
Heart rate | Continuous recording continuously throughout the 8-min exercise test using short-range radiotelemetry using a chest belt worn by the participant.
  Heart rate (beats per minute) will be recorded throughout the exercise challenge test to control intensity between trials.
Rating of breathing discomfort | Breathing discomfort severity ratings will be recorded every 2 minutes throughout the 8 min exercise test (a total of 4 measurements)
  Modified Borg scale (0- no discomfort, 10- severe discomfort).
Description of breathing discomfort | A description of breathing discomfort will be recorded every 2 minutes throughout the 8 min exercise test (a total of 4 measurements)
  Descriptors from patients to describe the level of discomfort - i.e. 'my chest is tight'.

CONTACTS AND LOCATIONS:
Overall Officials: Hannah Marshall, MSc, Principal Investigator — Brunel University
Locations (1):
- Brunel University London, Uxbridge, Middlesex, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided